CLINICAL TRIAL: NCT03704844
Title: Evaluation of the Renal Congestion, Perfusion and Function Before and After Diuretic Treatment in the ICU
Acronym: ECHOFURO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7148
Record Dates: First submitted 2018-07-30; First posted 2018-10-15 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Renal Congestion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with renal congestion
  Interventions: Other: non applicable
- Patients without renal congestion
  Interventions: Other: non applicable

INTERVENTIONS:
Other: non applicable — non applicable

SUMMARY:
Renal congestion is a pathological state that can lead to acute kidney failure. Furosemide is known to lower renal congestion by its diuretic effect.

The aim of this trial is to study the reversibility of kidney congestion under diuretic therapy and assess through echodoppler parameters if it can improve renal perfusion and function in congestive ICU patients.

It could in fine lead to a better identification of patients that could benefit from diuretic therapy in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in ICU
* under furosemide treatment

Exclusion Criteria:

* participation refusal
* uncontrolled shock (MAP<65mmHg)
* abdominal compartment syndrome
* diuretic administration in the 6 hours prior to inclusion
* renal replacement therapy or stage 4-5 chronic kidney disease
* atrial fibrillation
* no monitoring of CVP / invasive arterial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients under treatment by furosemide
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Effects of diuretics | 24 hours
  Evaluation of renal perfusion diuretic treatment by measuring the renal resistance index and the renal venous impedance index.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Amiens-Picardie, Amiens
  - CHU de Dijon, Dijon
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided